CLINICAL TRIAL: NCT05762250
Title: Auricular Acupuncture in Patients With Advanced Cancer: a Randomized Clinical Trial.
Acronym: MY_ACU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S00776
Record Dates: First submitted 2023-02-22; First posted 2023-03-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Fatigue; Pain; Depression; Advanced Tumour Diseases
Keywords: Auricular Acupuncture; advanced tumour diseases
MeSH Terms: conditions — Fatigue; Pain; Depression | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auricular Acupuncture (Experimental): Intervention group: Ear acupressure is performed on both ears with permanent pellets according to the NADA (National Acupuncture Detoxification Association) protocol over a period of 8 weeks (presentation at the study center 1x/week, application of the acupressure patches there; these remain on both ears for 5 days and should be massaged 3x/day by the patients themselves according to the instructions provided).
  In addition, patients receive a 30-minute psychoeducational talk at the first treatment appointment to promote their own health competence.
  Interventions: Other: Auricular Acupuncture
- Waitlist (No Intervention): Control group: standard treatment / waiting list Patients in the control group will also receive a one-time 30-minute psychoeducational interview at baseline.

INTERVENTIONS:
Other: Auricular Acupuncture — Within the NADA protocol, 5 defined points on the patient's ears are treated according to a standardized concept (shen men, kidney, lung, liver, vegetative I).
  Arms: Auricular Acupuncture

SUMMARY:
In the present study, the effect of ear acupressure treatment according to the NADA protocol on the quality of life of patients with advanced tumour diseases. (all stages) will be investigated. Furthermore, the effect of ear acupressure on anxiety and depression, pain, fatigue and sleep of the patients will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with advanced tumour diseases on current therapy, who suffer from persistent disease- or therapy-associated symptoms and limitations (screening by distress thermometer, score ≥ 5)
* Informed consent.

Exclusion Criteria:

* medical reasons or
* a mental condition which, in the opinion of the investigator, does not allow the patient to participate in the study,
* a planned radiation therapy in the area of the skull (to avoid potential scattered radiation),
* a missing legally binding signature on the informed consent form,
* participation in another acupuncture/acupressure study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-08-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in disease-specific quality of life (FACT-MM) | after 8 weeks (end of intervention)
  The FACT-MM can depict a more comprehensive picture of the patient's health status and collects data on precisely those areas that are most important to the patient himself.
  The diagnosis-specific subscale developed in this process assesses pain, fatigue, physical activity, emotional health, and cognitive abilities and represents the primary outcome parameter in this study.

SECONDARY OUTCOMES:
Change in anxiety and depressiveness | fourth week of intervention
  The four-item PHQ-4 is part of the PHQ-D, a health questionnaire for patients, and is composed of the PHQ-2, a two-item depression scale, and the GAD-2, a two-item anxiety scale.
Change in anxiety and depressiveness | after 8 weeks (end of intervention)
  The four-item PHQ-4 is part of the PHQ-D, a health questionnaire for patients, and is composed of the PHQ-2, a two-item depression scale, and the GAD-2, a two-item anxiety scale.
Change in anxiety and depressiveness | 2 weeks post-intervention
  The four-item PHQ-4 is part of the PHQ-D, a health questionnaire for patients, and is composed of the PHQ-2, a two-item depression scale, and the GAD-2, a two-item anxiety scale.
Change in anxiety and depressiveness | 12 weeks post-intervention
  The four-item PHQ-4 is part of the PHQ-D, a health questionnaire for patients, and is composed of the PHQ-2, a two-item depression scale, and the GAD-2, a two-item anxiety scale.
Change of individual symptom burden | fourth week of intervention
  Individual symptom burden - patients are asked to rate their 3 most distressing symptoms on a Numerical Rating Scale.
Change of individual symptom burden | after 8 weeks (end of intervention)
  Individual symptom burden - patients are asked to rate their 3 most distressing symptoms on a Numerical Rating Scale.
Change of pain | fourth week of intervention
  Improvement of pain (FACT-MM) questionnaire
Change of pain | after 8 weeks (end of intervention)
  Improvement of pain (FACT-MM) questionnaire
Change of pain | 2 weeks post-intervention
  Improvement of pain (FACT-MM) questionnaire
Change of pain | 12 weeks post-intervention
  Improvement of pain (FACT-MM) questionnaire
Change of Fatigue | fourth week of intervention
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item questionnaire designed to assess self-reported fatigue and its impact on daily activities and functions.
Change of Fatigue | after 8 weeks (end of intervention)
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item questionnaire designed to assess self-reported fatigue and its impact on daily activities and functions.
Change of Fatigue | 2 weeks post-intervention
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item questionnaire designed to assess self-reported fatigue and its impact on daily activities and functions.
Change of Fatigue | 12 weeks post-intervention
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13-item questionnaire designed to assess self-reported fatigue and its impact on daily activities and functions.
Change of sleep disorders and sleep quality | fourth week of intervention
  The Pittsburgh Sleep Quality Index (PSQI) was developed as a standardized self-assessment questionnaire by the University of Pittsburgh to elicit quality of sleep using qualitative and quantitative questions at a 4-week interval
Change of sleep disorders and sleep quality | after 8 weeks (end of intervention)
  The Pittsburgh Sleep Quality Index (PSQI) was developed as a standardized self-assessment questionnaire by the University of Pittsburgh to elicit quality of sleep using qualitative and quantitative questions at a 4-week interval
Change of sleep disorders and sleep quality | 2 weeks post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) was developed as a standardized self-assessment questionnaire by the University of Pittsburgh to elicit quality of sleep using qualitative and quantitative questions at a 4-week interval
Change of sleep disorders and sleep quality | 12 weeks post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) was developed as a standardized self-assessment questionnaire by the University of Pittsburgh to elicit quality of sleep using qualitative and quantitative questions at a 4-week interval
Number of pateints with adverse events | through study completion, an average of 3 Years
  Tolerability of the application

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Loeffler, Dr, Principal Investigator — University Hospital Wuerzburg
Locations (2):
- Germany (2):
  - Robert Bosch Krankenhaus, Stuttgart
  - University Hospital Wuerzburg, Würzburg